CLINICAL TRIAL: NCT02896036
Title: Laparoscopic Entry Technique With a Veress Needle Insertion With and Without Concomitant CO2 Insufflation - Does it Matter?
Brief Title: Veress Entry With/Without Concomitant CO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00025352
Record Dates: First submitted 2016-05-31; First posted 2016-09-12 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Laparoscopy; Laparoscopic Surgery; Insufflation; Gynecologic Surgical Procedures
Keywords: Laparoscopic Entry; Veress Needle; Intraperitoneal insufflation; Time; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Veress needle entry with concomitant CO2 (Experimental): For the group of participants who will be randomized to concomitant CO2 insufflation; the Veress will be connected to the CO2 tubing, and a skin incision will be made with the scalpel, followed by starting the CO2 gas insufflation and insertion of the Veress needle. If the opening pressure is less than or equal to 10 mmHg, the process of insufflation will be allowed to continue. In case of a higher opening pressure, the veress will be withdrawn and reinserted up to 3 times. A failed entry will be called if the peritoneal cavity cannot be insufflated after 3 attempts.
  Interventions: Procedure: Veress needle entry with concomitant CO2
- Veress needle entry with subsequent CO2 (Active Comparator): For the other group of participants who will be randomized to subsequent CO2 insufflation; the Veress needle will be connected to the CO2 tubing, and a skin incision will be made with the scalpel, followed by insertion of the Veress needle. The gas insufflation will be started and the opening pressure will be noted. If the opening pressure is less than or equal to 10 mmHg, the process of insufflation will be allowed to continue. In case of a higher opening pressure, the Veress needle will be withdrawn and reinserted up to 3 times. Each time the needle is to reinserted, the CO2 insufflator will be switched off until the location of the Veress needle is felt to be adequate.
  Interventions: Procedure: Veress needle entry with subsequent CO2

INTERVENTIONS:
Procedure: Veress needle entry with concomitant CO2 — The Veress will be connected to the CO2 tubing, and a skin incision will be made with the scalpel, followed by starting the CO2 gas insufflation and insertion of the Veress needle.
  Arms: Veress needle entry with concomitant CO2
Procedure: Veress needle entry with subsequent CO2 — A skin incision will be made with the scalpel. The Veress needle will be inserted until intraperitoneal location obtained. This will be followed by starting CO2 gas insufflation until the standard 15 mmHg.
  Arms: Veress needle entry with subsequent CO2

SUMMARY:
Purpose: The primary objective is to compare the time required for adequate intraperitoneal insufflation (from skin incision to reaching intraperitoneal pressure of 15 mmHg). Also the number of attempts needed before successful entry is achieved. The secondary objectives will evaluate rates of secondary outcomes measures such as; failed entry, extra peritoneal insufflation, vascular injury, visceral injury, gas embolism, solid organ injury, and omental injury between the two techniques.

Study design: prospective randomized control trial

Hypothesis: The investigators hypothesize that participant's undergoing laparoscopic surgery for benign Gynecologic indications at TGH who undergo laparoscopic entry technique of Veress needle entry with concomitant CO2 insufflation will require less time to achieve a 15 mmHg of intraperitoneal pressure as opposed to Veress needle entry with subsequent CO2 insufflation, and will require less number of attempts to achieve successful entry.

DETAILED DESCRIPTION:
Subject Recruitment and Consent:

All female patients age 18-70 scheduled for benign gynecologic laparoscopic surgery at TGH by a participating attending surgeon will be recruited. Each participant will be educated about the study; its objectives, potential benefits and risks, and the research team will obtain informed consent. Plan to enroll 90 participants.

Materials and Methods:

This will be a randomized control trial in which participants will be randomly assigned to have laparoscopic entry with Veress needle connected to CO2 tubing for concomitant insufflation versus Veress needle entry with subsequent connection to CO2 tubing for insufflation. The investigators will inform the patients about the two entry techniques during the pre-operative office visit. Participants will be consented to participate in the study prior to the surgery by the study research coordinators during their pre-operative visit. Patients who do not consent for the study will still undergo the scheduled procedure with standard entry technique as clinically indicated by their provider. Randomization will occur in the operating room just before the surgery starts. The healthcare provider performing the procedure will open the next sequentially numbered envelope, within which there will be a piece of paper indicating the entry technique to be performed. This will then be recorded in the study log. The study log will include enrolled participants, assigned study number which will range from 001 to the minimum number of participants required for the study as indicated by sample size calculation (see below). The participant will be positioned in the dorsal lithotomy position and prepped and draped in the standard fashion. Preoperative antibiotics will be provided as per standard indication for the procedure. For the group of participants who will be randomized to concomitant CO2 insufflation; the Veress will be connected to the CO2 tubing, and a skin incision will be made with the scalpel, followed by starting the CO2 gas insufflation and insertion of the Veress needle. If the opening pressure is less than or equal to 10 mmHg, the process of insufflation will be allowed to continue. In case of a higher opening pressure, the Veress will be withdrawn and reinserted up to 3 times. A failed entry will be called if the peritoneal cavity cannot be insufflated after 3 attempts. For the other group of patients who will be randomized to subsequent CO2 insufflation; the Veress needle will be connected to the CO2 tubing, and a skin incision will be made with the scalpel, followed by insertion of the Veress needle. The gas insufflation will be started and the opening pressure will be noted. If the opening pressure is less than or equal to 10 mmHg, the process of insufflation will be allowed to continue. In case of a higher opening pressure, the Veress needle will be withdrawn and reinserted up to 3 times. Each time the needle is to reinserted, the CO2 insufflator will be switched off until the location of the Veress needle is felt to be adequate. The time will be recorded from incision to the time it takes to achieve intraperitoneal pressure of 15 mmHg. In addition to the above primary and secondary outcomes of the study, participant demographic information, procedure specific variables and outcomes will be collected and recorded in the study log (See data collection sheet). Common laparoscopic complications will also be recorded, including the following:

* Vascular injury: any tear or injury to any intraabdominal blood vessels.
* Visceral injury: any serosal (superficial) or full thickness (deep) injury to the small or the large bowel.
* Gas embolism: entrapment of carbon dioxide in an injured vein, artery or solid organ, and results in blockage of the right ventricle (RV) or pulmonary artery
* Solid organ injury: any injury of a solid abdominal or pelvic organ including but not limited to, liver, spleen or the uterus.
* Failed entry: failure to establish pneumoperitoneum after 3 attempts of Veress insufflation.
* Extraperitoneal insufflation: insufflating the preperitoneal space with carbon dioxide.
* Omental injury: any injury to the greater omentum that results in bleeding of omental insufflation.

Sample size: 90 patients will be recruited based on the sample size calculations already performed.

ELIGIBILITY:
Inclusion Criteria:

* All female patients within the ages of 18-70 presenting to TGH for benign gynecologic laparoscopic surgery performed by the study investigators. The following surgeries will be considered as part of the study:

  * Diagnostic laparoscopy
  * Laparoscopic adnexal surgery
  * Laparoscopic hysterectomy
  * Laparoscopic myomectomy
  * Robotic assisted hysterectomy
  * Robotic assisted myomectomy

Exclusion Criteria:

* Patients unable to provide informed consent
* Previous midline laparotomy
* 3 or more previous cesarean sections through a Pfannenstiel incision

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Time required for adequate intraperitoneal insufflation. | intraoperative
  Time from insertion of Veress to insufflation of peritoneum to 15 mmHg.

SECONDARY OUTCOMES:
Evaluate rates of failed entry between the two techniques | intraoperative
  Evaluate occurrence of failed entry (more than 3 attempts with the Veress without intraperitoneal insufflation)
Evaluate rates of extraperitoneal insufflation between the two techniques | intraoperative
Evaluate rates of vascular injury between the two techniques | intraoperative
Evaluate rates of visceral injury between the two techniques | intraoperative
Evaluate rates of gas embolism between the two techniques | intraoperative
  omental injury between the two techniques
Evaluate rates of solid organ injury between the two techniques | intraoperative
Evaluate rates of omental injury between the two techniques | intraoperative
Evaluate number of entry attempts. | intraoperative
  Record the number of attempts taken with Veress needle to obtain successful intraperitoneal entry.

CONTACTS AND LOCATIONS:
Overall Officials: Emad Mikhail, MD, Principal Investigator — University of South Florida Department of Obstetrics and Gynecology; Anthony Imudia, MD, Study Director — University of South Florida Department of Obstetrics and Gynecology; Elisabeth Sappenfield, MD, Study Chair — University of South Florida Department of Obstetrics and Gynecology
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No